CLINICAL TRIAL: NCT00284726
Title: A Prospective, Controlled, Randomized Study on the Effect of Cold Storage Solutions on Complement Activation and Other Mediators of Ischemic Injury in Lung Transplantation
Brief Title: The Effect of Cold Storage Solutions on Ischemic Injury in Lung Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Other Study IDs: 00-10-25-03
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2017-12

CONDITIONS: Lung Transplant Recipients
Keywords: Cytokines in lung transplantation; Cold storage solutions; Ischemic reperfusion injury

INTERVENTIONS:
Device: Celsior Cold Storage Solution

SUMMARY:
The purpose of this study is to compare 2 different cold storage solutions, used to preserve donor lungs for lung transplantation, and their effect on cytokine activation related to ischemic reperfusion injury. Primary endpoint is 30 day survival.

DETAILED DESCRIPTION:
The length of ischemic time in harvesting lung allografts is associated with graft survival. It is further thought that ischemic changes in early post-transplantation bronchoscopic biopsies has a direct correlation with later development of chronic rejection.

ELIGIBILITY:
Inclusion Criteria:

Any patient undergoing a lung trasnplant at Johns Hopkins Hospital -

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-12; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: John V. Conte, M.D., Principal Investigator — Johns Hopkins University